CLINICAL TRIAL: NCT07388368
Title: A Comparative Evaluation of Post Obturation Pain After Root Canal Treatment Using Tricalcium Silicate Versus Resin-based Sealers in Cases With Symptomatic Irreversible Pulpitis
Brief Title: Comparative Evaluation of Post Obturation Pain After Root Canal Treatment Using Tricalcium Silicate vs Resin-Based Sealers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Pooja Kumari, Dr. Pooja Kumari, Principal Investigator and Resident, Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol-001
Record Dates: First submitted 2025-12-07; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: root canal sealar; postobturation pain; bioceramic sealer; resin based sealar
MeSH Terms: conditions — Pain | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Intervention Model Description: A comparative evaluation of postobturation pain after root canal treatment using tricalcium silicate versus resin-based sealers in cases with symptomatic irreversible pulpitis
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tricalcium silicate based sealer (Bio ceramic) (Active Comparator): CeraSeal bioceramic sealer will be used for obturation with matched bioceramic cones and a heated plugger (System B).
  Interventions: Drug: Tricalcium silicate sealar
- Resin based sealer (Experimental): Endoplus resin-based sealer will be used for obturation with single-cone gutta-percha and a heated plugger (System B)
  Interventions: Drug: Resin based sealer

INTERVENTIONS:
Drug: Tricalcium silicate sealar — Ceraseal (bioceramic sealer) - assigned to Group 2
  Other Names: CeraSeal sealer, bioceramic sealer, calcium silicate sealer
  Arms: Tricalcium silicate based sealer (Bio ceramic)
Drug: Resin based sealer — Endoplus (resin-based sealer) - assigned to Group 1
  Other Names: Endoplus sealer, resin sealer, gutta-percha sealer
  Arms: Resin based sealer

SUMMARY:
This is a randomized controlled trial comparing the mean and standard deviation of postobturation pain using two different sealers: a tricalcium silicate-based sealer (CeraSeal) and a resin-based sealer (Endoplus) in patients with symptomatic irreversible pulpitis undergoing root canal treatment.

DETAILED DESCRIPTION:
• The study will be conducted after approval from the Institutional Ethics Review Committee of the Armed Forces Institute of Dentistry. Informed written consent will be obtained from all patients, and demographic details (name, age, gender, and contact information) will be collected. This is a randomized clinical trial, and the sample size will be divided into two groups using computer-generated randomization. Group 1 will receive Endoplus (resin-based sealer), and Group 2 will receive CeraSeal (bioceramic sealer).

All root canal procedures will be performed by the principal investigator. At the first visit, local anesthesia (2% lignocaine with 1:100,000 epinephrine) and rubber dam isolation will be used. Working length will be determined using an apex locator and confirmed with a periapical radiograph. Chemo-mechanical preparation will be performed using 2.5% sodium hypochlorite (NaOCl) and 17% ethylenediaminetetraacetic acid (EDTA). Cleaning and shaping will be done up to F2 ProTaper using hand files and nickel-titanium (NiTi) rotary files, with recapitulation between each file to maintain canal patency. Non-setting calcium hydroxide will be placed as an intracanal medicament, followed by a temporary restoration with Cavit. Patients will be recalled after one week for obturation and will proceed only if asymptomatic.

At the second visit, obturation will be carried out according to group allocation. Group 1 will receive Endoplus resin-based sealer using a single-cone gutta-percha technique with a heated plugger (System B). Group 2 will receive CeraSeal bioceramic sealer with matched bioceramic cones using the same System B technique. Accessory cones will be used for wide or irregular canals. A permanent composite restoration (Coltene) will be placed, and occlusion will be adjusted.

Postoperative pain will be recorded using a Visual Analogue Scale (VAS) at 24 hours, 72 hours, and 7 days. Ibuprofen will be prescribed only if the pain becomes unbearable, and patients will document the dose and frequency taken. Two independent blinded endodontists will evaluate radiographs for technical errors or sealer extrusion. The primary measure of success will be the level of postoperative pain at follow-up, comparing outcomes between Endoplus resin-based sealer and CeraSeal bioceramic sealer.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of age group 18 to 60 years

  * Healthy patients with ASA class 1 and 2
  * Patients of both genders
  * Teeth diagnosed as symptomatic irreversible pulpitis
  * Single as well as multirooted teeth

Exclusion Criteria:

* Teeth with calcified or previously treated canals
* Immunocompromised or mentally handicapped patients
* Pregnant or lactating mothers
* Teeth with periodontal probing depths of 5 mm or more
* Cracked or un restorable teeth
* Teeth where root canal instrumentation could not reach within 2 mm of the radiographic apex

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain after root canal treatment assessed using a Visual Analogue Scale (VAS) | 24 hours, 72 hours and 7 days
  Postoperative pain will be recorded using a 10-centimeter Visual Analogue Scale (VAS). On this scale, 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores correspond to greater pain intensity, meaning more pain. Patients will self-report their pain level at each time point (24 hours, 72 hours, and 7 days). This measure will be used to compare postoperative pain between patients treated with Endoplus resin-based sealer and CeraSeal bioceramic sealer.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Force Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers because this trial involves a small patient sample, and the data contains identifiable clinical information that cannot be fully anonymized without compromising patient confidentiality. The dataset is intended solely for analysis within the approved research protocol, as permitted by the Institutional Ethics Review Committee. Therefore, IPD sharing is not planned.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT07388368/Prot_SAP_ICF_000.pdf